CLINICAL TRIAL: NCT01426932
Title: The Head Impulse Test in the Screening of Vestibular Function
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services, Haifa and West Galilee (Other)
Responsible Party: Sponsor
Other Study IDs: HITVNG
Record Dates: First submitted 2011-08-27; First posted 2011-09-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2012-02

CONDITIONS: Vertigo
Keywords: Vestibular Function Tests; Caloric Test; Electronystagmography; Prediction
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Video recording of Head Impulse Test — Video recording of Head Impulse Test

SUMMARY:
The alternate binaural bithermal caloric test (ABBT) is a well established examination in the evaluation of the dizzy patient. ABBT is useful in detecting the side of peripheral vestibulopathy by stimulating each ear separately, it contributes to the diagnosis of bilateral vestibular involvement when all responses to cold and warm stimuli are reduced, and adds to the differentiation of peripheral from central vestibular involvement by measuring the fixation-induced inhibition of the caloric response. In spite of these benefits, ABBT is the most time-consuming part of the electronystagmography/Videonystagmography (ENG/VNG) test battery, and frequently causes significant inconvenience to the patient due to the repeated extreme vestibular stimuli.

The head impulse test (HIT) assesses vestibular function by brisk, passive rotations of the head in the plane of the examined semicircular canals. Whenever the vestibulo-ocular reflex (VOR) is deficient, this maneuver would produce catch-up saccades aiming to the re-fixation of the eyes on the target. Hence, both residual VOR and catch-up saccades act synergistically to stabilize gaze. The HIT requires only several minutes and might cause minimal discomfort only.

The study hypothesis is that the HIT recorded by standard VNG equipment of the VNG system would provide diagnostic information on the side of vestibular involvement matching that of the ABBT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Videonystagmography(VNG) test battery is indicated for the diagnosis of dizziness or vertigo

Exclusion Criteria:

* Signs of retrocochlear lesion or central vestibular pathology in bed-side otoneurological examination or audiometry or ENG/VNG
* Age < 18 years
* Otitis externa
* Otitis media
* Tympanic membrane perforation
* Status Post Mastoidectomy
* Limitations of neck movements in the horizontal plain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary center patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the recorded HIT results in the prediction of the caloric test lateralization parameter | 18 months
  Sensitivity would be calculated according to the following formula: Number of participants in whom catch-up saccades would be recorded and caloric test lateralization would be greater than 25% divided by the sum of number of participants in whom catch-up saccades would be recorded and caloric test lateralization would be greater than 25% plus the number of participants in whom no catch-up saccades would be recorded and caloric test lateralization would be greater than 25% (number of true positives /(number of true positives + number of false negatives))
Specificity of the VNG recorded HIT results in the prediction of the caloric test lateralization parameter | 18 months
  Specificity would be calculated according to the following formula: Number of participants in whom no catch-up saccades would be recorded and caloric test lateralization would be smaller than 25% divided by the sum of number of participants in whom no catch-up saccades would be recorded and caloric test lateralization would be smaller than 25% plus the number of participants in whom catch-up saccades would be recorded and caloric test lateralization would be smaller than 25% (number of true negatives /(number of true negatives + number of false positives))

SECONDARY OUTCOMES:
Sensitivity of the bed-side HIT examination results in the prediction of the caloric test lateralization parameter | 18 months
  Sensitivity = Number of participants in whom catch-up saccades would be diagnosed in the HIT bed-side examination and caloric test lateralization would be greater than 25% divided by the sum of number of participants in whom catch-up saccades would be diagnosed in the HIT bed-side examination and caloric test lateralization would be greater than 25% plus the number of participants in whom no catch-up saccades would be diagnosed and caloric test lateralization would be greater than 25% (number of true positives /(number of true positives +number of false negatives))
Specificity of the bed-side HIT examination results in the prediction of the caloric test lateralization parameter | 18 months
  Specificity would be calculated according to the following formula: Number of participants with no catch-up saccades in the HIT bed-side examination and caloric test lateralization smaller than 25% divided by the sum of number of participants in with catch-up saccades in the HIT bed-side examination and caloric test lateralization smaller than 25% plus the number of participants with catch-up saccades in the HIT bed-side examination and caloric test lateralization smaller than 25% (number of true negatives /(number of true negatives + number of false positives))

CONTACTS AND LOCATIONS:
Locations (1):
- Otoneurology Unit, Lin Medical Center, 35 Rotchild Avenue, Haifa, Israel